CLINICAL TRIAL: NCT06629792
Title: A Clinical Study To Evaluate the Efficacy and Tolerance of a Topical Facial Treatment on Women With Mild to Moderate Fine Lines, Wrinkles, and Laxity on the Global Face
Brief Title: A Clinical Study Evaluating the Efficacy and Tolerability of a Topical Facial Treatment For Facial Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Revision Skincare (Industry)
Collaborators: SGS Stephens, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C22-D008
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Fine Lines; Wrinkles; Laxity; Skin
Keywords: topical treatment; skin rejuvenation; anti-aging
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Topical Treatment (Experimental): Subjects received a topical facial treatment applied by a license esthetician in a series of 3 sessions at 1 month intervals, in combination with a cleanser, moisturizer, and sunscreen over the course of 12 weeks.
  Interventions: Other: Gentle Cleanser; Other: Facial Moisturizer; Other: sunscreen SPF 30

INTERVENTIONS:
Other: Gentle Cleanser — The cleanser was instructed to be used twice daily over the course of 12 weeks
  Other Names: Gentle Foaming Cleanser, Revision Skincare
Other: Facial Moisturizer — The Moisturizer was instructed to be applied to the global face twice daily over the course of 12 weeks.
Other: sunscreen SPF 30 — The Sunscreen was instructed to be applied once daily in the morning, with re-application with extended sun exposure per FDA guidelines over the course of 12 weeks.
  Other Names: Neutrogena Ultra Sheer Dry-Touch Sunscreen SPF 30

SUMMARY:
This single-center clinical trial was conducted to evaluate the efficacy and tolerability of a topical facial treatment when applied by a license esthetician in clinic in a series of 3 sessions with 1 month intervals, in combination with a cleanser, moisturizer, and sunscreen over the course of 12 weeks in healthy women aged 35 to 60 with mild to moderate global facial fine lines, wrinkles, and laxity. Thirty-two (32) healthy female subjects completed the clinical study.

DETAILED DESCRIPTION:
This single-center clinical trial was conducted to evaluate the efficacy and tolerability of a topical facial treatment when applied by a license esthetician in clinic in a series of 3 sessions with 1 month intervals, in combination with a cleanser, moisturizer, and sunscreen over the course of 12 weeks in healthy women aged 35 to 60 with mild to moderate global facial fine lines, wrinkles, and laxity.

The efficacy and tolerability of the topical facial treatment in improving mild to moderate global facial fine lines, wrinkles, and laxity. was evaluated by Investigator clinical efficacy grading and tolerability grading by a board-certified dermatologist, subject tolerability grading, and clinical photography.

ELIGIBILITY:
Inclusion Criteria:

* Having Fitzpatrick Skin Type I - VI
* Having mid to moderate global face fine lines, wrinkles, and laxtiy (tactile) (score of 3 to 6 according to a modified Griffiths scale).

Exclusion Criteria:

* Breastfeeding, pregnant, or planning to become pregnant during the study.
* Currently having or having a history of cold sores (Herpes simplex) on the face.

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Change Investigator Clinical Efficacy Grading versus Baseline | 12 weeks
  The primary efficacy endpoint will be Investigator Clinical Efficacy grading of parameters at baseline, post-application, and weeks 4, 8, and 12. the efficacy parameters will be assessed by the expert grader on each subjects global face using a modified Griffiths 10-point scale. A decrease in score indicates an improvement.
Lack of significant change in Investigator Tolerability Parameters versus Baseline | 12 weeks
  The primary tolerability endpoint will be Investigator Tolerability Assessment of at baseline, post-application, and weeks 4, 8, and 12. Local cutaneous tolerability will be evaluated by the expert grader by assessing the signs of erythema and dryness using a four-point scale: 0 = None 1 = Mild 2 = Moderate 3 = Severe. A decrease in score indicates an improvement.
Lack of significant change in Subjective Tolerability versus Baseline | 12 weeks
  The primary tolerability endpoint will be Subjective Tolerability Assessment of at baseline, post-application, and weeks 4, 8, and 12. Local cutaneous tolerability will be evaluated by subject reporting of the degree of burning, stinging, and itching globally on each subject's global face using a four-point scale: 0 = None 1 = Mild 2 = Moderate 3 = Severe. A decrease in score indicates an improvement.

SECONDARY OUTCOMES:
Change in Facial Parameters in a Self-Assessment Questionnaire versus Baseline and Percent Agreement | 12 weeks
  The secondary endpoint will be subject self-assessment questionnaire completed at baseline, post-application, and weeks 4, 8, and 12. Subjects are asked to rate statements based on a scoring system ranging from 5 (completely agree) to 1 (completely disagree). A change in response values at post-application, and weeks 4, 8, and 12 compared to baseline response values indicates an improvement. The best outcome is to Completely Agree with the statement / question being asked.
Clinical Photography: VISIA-CR and Antera 3D | 12 weeks
  The secondary endpoint will be image analysis of VISIA-CR and Antera 3D clinical photography. VISIA-CR imaging analysis for nasolabial folds, and Antera imaging analysis of roughness and volume on images taken at all timepoints. a reduction in visual fine lines, wrinkles, radiance, and laxity on post-baseline timepoints compared to baseline is indicated an improvement

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Stephens, inc., Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: No